CLINICAL TRIAL: NCT01569555
Title: Crossed Leg Sign and it's Correlation With Significant Pathology
Brief Title: Significant Pathology Associated With Crossed Leg Sign
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uelk, J. Daniel, D.O. (Individual)
Responsible Party: Sponsor
Other Study IDs: 7286
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: Pathology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
By determining the correlation of a Crossed Leg Sign with signifcant pathology, a clinician would then be able to use this correlation to risk stratify his/her patients for significant pathology.

DETAILED DESCRIPTION:
By determining the correlation of a Crossed Leg Sign with signifcant pathology, a clinician would then be able to use this correlation to risk stratify his/her patients for significant pathology. Therefore, by determining the sensitivity and specificity of this physical exam finding, the clinician would have a better idea of the patients clinical management, including diagnostic testing and ultimate treatment of the patient. Crossed Leg Sign will be defined in this study as: any patient observed in the Emergency Department with sustained crossed legs. To my knowledge, crossed legs have never been evaluated in regards to it's correlation with significant pathology. This could potentially add another physical exam finding to be used by the clinician.

ELIGIBILITY:
Inclusion Criteria:

* Any patient observed in the Emergency Department with sustained crossed legs.

Exclusion Criteria:

* Any patient not observed to have sustained crossed legs and is not being used as a control.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study should include all comers. To exclude a patient population would add a selection bias.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John D Uelk, DO, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Wyandotte Hospital, Wyandotte, Michigan, United States